CLINICAL TRIAL: NCT06259305
Title: Study of the Feasibility and Acceptability of Using Antenatal Music Therapy for Families Experiencing Pregnancies Where the Foetus Has a Life-Limiting Diagnosis
Brief Title: Memories in Heartbeats Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UHDB/2022/087S
Record Dates: First submitted 2023-08-23; First posted 2024-02-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-04

CONDITIONS: Palliative Care
Keywords: Palliative Care; Pregnancy

STUDY DESIGN:
Intervention Model Description: Observational,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Creation of a memory track combined with the baby's heartbeat (Experimental): A memory track will be created by the music therapist with the family and this will be overlaid with a recording of the baby's heartbeat, provided by the family.
  This recording will be placed inside a memory bear and given to the family to keep.
  This will be offered to form part of the memory making process alongside existing processes.
  Interventions: Other: Creation of a memory track combined with the baby's heartbeat

INTERVENTIONS:
Other: Creation of a memory track combined with the baby's heartbeat — This is as described above

SUMMARY:
A small feasibility study to explore the role of music therapy as part of memory making experiences in mothers who are experiencing a pregnancy where screening tests show that the foetus has a condition meaning they may not develop to full term, survive the birth or that the new-born will have continued complications and limited life expectancy once born. The outcome of this study will be to determine the feasibility and acceptability of offering antenatal music therapy for families experiencing pregnancies where a foetal condition or anomaly means that comfort care only is planned for the baby after birth and to assess if the development of a musical memory-making tool will be relevant for this patient group within the current bereavement midwifery services. The study plans to use the recorded heartbeat of the unborn foetus and then to combine this with music of the family's choice to create a memory track which can then be saved into a recording device such as a memory bear for the family to keep. It is proposed that this intervention could complement current memory making processes already being offered by services such as bereavement midwives working within Hospital trusts.

DETAILED DESCRIPTION:
It is evident from research that music, and in particular music therapy, can be hugely beneficial throughout pregnancy for both a mother and her developing baby (Lander, 2017; Arya et al, 2012). Communication, building relationships and relaxation are just some of the benefits experienced during the antenatal period and can be linked with postnatal experiences and development, in particular, within the Neonatal Intensive Care Units (NICUs) (Keith, Russell & Weaver, 2009, Ettenberger, 2017, Roa & Ettenberger, 2018).

However, comprehensive literature reveals little evidence about music therapy in pregnancies where screening tests show the foetus has a condition meaning they may not develop to full term, survive the birth or that the newborn will have ongoing complications and limited life expectancy. Having this knowledge and deciding to continue with the pregnancy undoubtedly has an impact on the antenatal bonding process and finding ways to connect with "the bump" are incredibly important (Mastnak, 2016).

This study proposes to explore the role music therapy can play in antenatal bonding and memory making experiences prior to birth. This uses recordings of the baby's heartbeat combined with precomposed music to create a memory track which can then be saved into a recording device such as a memory bear.

The study will involve a single recruiting site, the Rainbows Hospice for Babies, Children and Young Adults where the Principal Investigator (PI) is the music therapist who will undertake all the study procedures with the participants.

The two NHS Trusts (University Hospitals of Derby and Burton NHS Trust and Leicester University Hospitals) will be participant identification centres (PICs). Potential participants will be identified by the clinical staff delivering usual clinical care. They will then make the first approach and if the potential participant is interested, give them a Participant Information Sheet (PIS). The PIS will contain the contact details for the PI. The potential participant may contact the PI directly if they are interested in discussing the study further or participating.

Due to limited time available, the time between identification of the potential participant and consent may be short but there will be no pressure to make a decision. Participants will take as long as they wish to make this decision, in line with their clinical care and the usual clinical care and referral pathways will not be affected by this process.

If the potential participant wishes to participate, they will be invited to meet the PI, discuss any further questions about the study and will be asked to grant written informed consent. Following consent, minimal demographic and clinical information will be recorded and an appointment made to complete the intervention visit and this is the stage at which participants will be asked to share the recording of baby's heartbeat with the researcher. The visit will also include a discussion to understand what music, nursery rhyme, or other type of recording the family would like to use with the heartbeat. These will be facilitated by the PI who is an experienced music therapist. The music therapy intervention session will last between 1-2 hours and the part that will be used in the memory making will be audio recorded. The completed recording will be shared with the family and will be offered to the family in their preferred format such as being placed inside a "memory bear".

Following this, the participant will be invited to the post-intervention interview 6 months later. The interview will be offered as face to face but could be by telephone/web-based if the participant prefers. This will be a semi-structured interview, which will be audio-recorded, and will explore the acceptability of the intervention and the participant experience using a topic guide. If the participants want to know and have given written consent for it, the results of the study will be communicated to them.

ELIGIBILITY:
Inclusion Criteria:

* · Pregnant people aged 18 and over

  * Experiencing a pregnancy where, due to a foetal diagnosis, the baby is unlikely to survive to full term or a comfort care only plan for postnatal care has been agreed between the parents and the health care professionals
  * Subjects capable of giving informed consent
  * Subjects have sufficient comprehension of the English language to enable informed consent
  * Subjects have, or can get, a recording of their baby's heartbeat that they are willing to share with the PI for the purpose of the study

Exclusion Criteria:

* · Pregnant people <18 years of age

  * Lack of capacity to provide informed consent
  * Have insufficient comprehension of the English Language to provide informed consent
  * No recording of baby's heartbeat, and not able to get one, or not willing to share with the PI for the purpose of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who will give consent for participation | 1 year
  Number of participants who will give consent for participation
Number of participants who complete music therapy | 1 year
  Number of participants who complete music therapy

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Ojha, Study Director — University Hospitals of Derby and Burton NHS Trust
Locations (1):
- Rainbows Hospice for Babies, Children and Young Adults Rainbows will be will be undertaking some of the core study coordination/management activities, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on reasonable request to the Chief Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available from end of study to 5 years
Access Criteria: Data will be made available on reasonable request to the Chief Investigator. The data will be completely anonymised and de-identified in line with the study protocol.